CLINICAL TRIAL: NCT03288077
Title: Nutrients to Enhance Sleep Quality and Quantity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-1420
Record Dates: First submitted 2017-09-18; First posted 2017-09-19 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Sleepiness in Athletes
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triptophan beverage (Experimental): Proprietary blend of nutritional interventions aimed at increasing sleepiness
  Interventions: Other: Tryptophan

INTERVENTIONS:
Other: Tryptophan — Beverage including tryptophan

SUMMARY:
Identifying non-pharmacological means of enhancing sleep is an important area of research for elite athletes. Research completed at the AIS has identified that some athletes have difficulties falling and staying asleep during both training and competition.

There are a number of dietary components such as nutrients and certain dietary supplements that are purported to decrease sleep latency and increase quality of sleep. While many of these interventions have been investigated in isolation, no research has examined different combinations and/or amounts of these substances to determine the resultant effects on sleep. The results of such a systematic investigation could produce an effective diet based sleep product ("Sleep Drink').

The optimal components, amounts, and timing of intake of such a Sleep Drink will be explored. Additionally, the effects on sleep will be evaluated using the gold standard of sleep measurement: polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 year old males

Exclusion Criteria:

* Exclusion: Exclusion criteria will include any observed or disclosed injury, illness, sleep or health issue which may disrupt the subject's performance or endanger their health. Participants will need to complete an adult screening tool, as recommended by Exercise and Sports Science Australia (ESSA), to assess this.
* Blood samples will also be collected to screen for magnesium, zinc and B12 which may influence nutritional impact on sleep. If subjects score above the reference ranges for these measures, they will be excluded.
* The Pittsburg Sleep Quality Index (PSQI) and Stanford Sleepiness Scale (SSS) will be used to screen for sleep disturbances. If subjects score outside the reference ranges for these questionnaires, they will be excluded.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
polysomnography | 0-3 hours
  The effect of the drinks will be determined primarily by polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Shona Halson, PhD, Principal Investigator — AIS

IPD SHARING:
Plan to Share IPD: No